CLINICAL TRIAL: NCT00936754
Title: Safety and Efficacy of a Unique Dose of a Brown Seaweeds Powder Enriched in Polyphenols on Human
Brief Title: Safety and Efficacy of a Single Dose of a Polyphenol-enriched Brown Seaweed Powder in Human
Acronym: ICAST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: innoVactiv Inc. (Industry)
Responsible Party: Jocelyn Bérubé/Scientific Director, Health & Nutrition, innoVactiv inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2005-RD-10-CLN2
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Glycemic Index
Keywords: Glycemic index; Reduction of glycemic index of ingested foods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Single administration of 500 mg of encapsulated brown seaweed powder, taken 30 minutes before test meal
  Interventions: Dietary Supplement: Brown seaweed powder
- Placebo (Placebo Comparator): Single administration of encapsulated placebo, taken 30 minutes before test meal
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Brown seaweed powder — 500 mg (in two 250 mg capsules) taken with 250 ml of water 30 minutes before test meal (110g of plain white bread with 250 ml of water)
  Arms: Treatment
Dietary Supplement: Placebo — Two capsules similar in aspect and weight to active product, taken with 250 ml of water 30 minutes before test meal (110g of plain white bread with 250 ml of water)
  Arms: Placebo

SUMMARY:
The primary endpoint of this trial will be to evaluate the safety of a single administration in human of a dose of 500 mg of a polyphenol-rich algal powder when taken 30 minutes before a test meal. The secondary endpoint of this trial will be to evaluate if a single administration in human of a dose of 500 mg of a polyphenol-rich algal powder is able to reduce the rate of carbohydrate absorption as measured by following postprandial glycemia and insulinemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* BMI between 20 and 30
* Non-smoking

Exclusion Criteria:

* Iodine allergy
* Diabetes
* Use of dietary supplements for duration of study
* History of major surgeries or surgeries of the stomach or digestive tract

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety of a single 500 mg administration of a brown seaweed extract in human | First administration up to 7 days after last administration

SECONDARY OUTCOMES:
Significant reduction of glycemic index of test food | Immediately after product administration (single use)
Significant reduction in postprandial glycemia | Immediately after product administration (single use)
Significant reduction in postprandial insulinemia | Immediately after product administration (single use)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, Principal Investigator — Institut des nutraceutiques et des aliments fonctionnels
Locations (1):
- Institut des Nutraceutiques et des Aliments Fonctionnels (INAF), Québec, Quebec, Canada